CLINICAL TRIAL: NCT06050018
Title: Effect of Milk Consumption on Gut Microbiome and Bone Remodeling Assessed by Serum C-telopeptide (CTX), Osteocalcin (OC) and Parathyroid Hormone (PTH) in Postmenopausal Women
Brief Title: Milk on Gut Microbiome and Bone Remodeling CTX in Postmenopausal Women
Acronym: Milk-CTX-GM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel Aviv University (Other)
Collaborators: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Prof Daniela Jakubowicz MD, Tel Aviv University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0203-22 WOMC
Record Dates: First submitted 2023-09-08; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Menopause

STUDY DESIGN:
Intervention Model Description: In a crossover design the effect of Yes Milk Diet (YesMdiet) and of No Milk Diet (NoMdiet) on Gut Microbiome (GM) and Bone Turnover Markers will be assessed in the participants in random order
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YesMilkdiet (Experimental): After one week baseline, the participants will be assigned to YesMilkdiet consuming milk and dairy products for 4 weeks
  Interventions: Other: YesMilkdiet
- NoMilkdiet (Active Comparator): After one week baseline, the participants will be assigned to NoMilkdiet consuming another source of protein and without milk or dairy products for 4 weeks
  Interventions: Other: NoMilkdiet

INTERVENTIONS:
Other: YesMilkdiet — In the YesMilkdiet the participants will consume Milk and dairy products
  Other Names: YesMdiet
  Arms: YesMilkdiet
Other: NoMilkdiet — In the NoMilkdiet the participants will not consume milk or dairy products only another sources of proteins
  Other Names: NoMdiet
  Arms: NoMilkdiet

SUMMARY:
Milk consumption drives beneficial effect on Bone Mass Density and on Gut Microbiome. Altered Gut Microbiome is associated with postmenopausal status, reduced Bone Mass Density, abnormal serum levels of Bone Turnover Markers (BTM), and disrupted T-cell immune mediation of several proinflammatory cytokines. The investigators hypothesize that a dietary intervention supplemented with milk and other non-fermented dairy products (YesMdiet), compared to an isocaloric diet with equivalent protein and calcium content but non-dairy protein sources (NoMdiet), will lead to favorable changes of Gut Microbiome [Primary end-point] in association with improved serum Bone Turnover Markers and serum proinflammatory cytokine profiles.

DETAILED DESCRIPTION:
Milk consumption is associated with favorable effects on Bone Mass Density, prevention of osteoporosis and beneficial changes in Gut Microbiome. Alteration of Fecal or Gut Microbiome (dysbiosis) is related to disturbances of osteoblastic bone formation and osteoclastic resorption, reduced Bone Mass Density, and abnormal serum levels of Bone Turnover Markers including serum Cross Linking C-telopeptide of Type 1 Collagen (s-CTX) or C-terminal telopeptide (CTX).The mechanism behind the deleterious effect of abnormal Gut Microbiome (GM) composition on bone includes effects on gut permeability, reduced production of short chain fatty acids, reduced insulin-like growth factor-1 and disrupted serum levels of T-cell immune mediation of several proinflammatory cytokines, e.g. tumor necrosis factor α (TNFα), transforming growth factor beta (TGF beta) and interleukin-17 (IL-17).

The investigators hypothesize that a dietary intervention (DI) supplemented with milk and other non-fermented dairy products (YesMdiet), compared to an isocaloric diet with equivalent protein and calcium content but non-dairy protein sources i.e., calcium-fortified soy and tofu or cheese substitutes (NoMdiet), will lead to favorable changes in composition and diversity in fecal samples for GM [Primary end-point] in association with improved serum Bone Turnover Markers namely of serum C-terminal telopeptide (CTX). and in serum levels of proinflammatory cytokine profiles. The effect of the two DI on Gut Microbiome and Bone Turnover Markers will be assessed in a random cross-over design. The cohort will include 15 postmenopausal women. GM and serum Bone Turnover Marker C-terminal telopeptide (CTX), and serum proinflammatory cytokines, will be assessed before and after 4 weeks of each diet intervention, (YesMdiet and NoMdiet), separated by 2 weeks of washout. Gut Microbiome composition and diversity will be assessed in fecal samples using 16S ribosomal RNA (rRNA) gene sequencing and shotgun metagenomics. Serum levels of Bone Turnover Marker C-terminal telopeptide (CTX), and serum levels of proinflammatory cytokines including tumor necrosis factor α (TNFα), transforming growth factor β (TGFβ) and interleukin-17 (IL-17), will be assessed in fasting serum samples.

This study will reveal whether dairy consumption improves the Gut Microbiome profile as well as serum Bone Turnover Marker C-terminal telopeptide (CTX), and proinflammatory cytokines in post-menopausal women, and will help to assess its value of dairy consumption as a potential intervention tool for preserving Bone Density and management of osteoporosis in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal status, defined by ≥ 1 year since last menstrual period and/or serum FSH ≥ 30 IU/l
* Normal liver, thyroid, parathyroid and kidney function eGFR > 60ml/min
* Usual Milk and milk products consumption

Exclusion Criteria:

* Diabetes,
* Prior osteoporotic fracture
* eGFR <60ml/min.
* Vitamin D 25-OH deficiency <10 ng/ml.
* Hypercalcemia Ca > 11.
* Chronic gastrointestinal disease, or acute condition with nausea, vomiting or diarrhea in the past month.
* Bariatric Surgery.
* Known hypersensitivity to milk components or lactose intolerance.
* Vegan/vegetarian
* Treatment with antibiotics or ingestion of prebiotics or probiotics in the 3 months preceding the study.
* Use of anti-osteoporosis medicines (e.g., bisphosphonates, raloxifene, calcitonin, teriparatide, and denosumab) within 36 months before enrollment.
* Use of Hormone replacement therapy, Vitamin K antagonists (e.g., warfarin), heparin, thiazide diuretics, anticonvulsants, aromatase inhibitors.
* Illicit drug abuse or alcoholism within one year prior to study onset;
* Use of glucocorticoids within 3 months prior to study onset.

Ages: 48 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only menopausal women will be recruited
Enrollment: 15 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiome Profile | 4 weeks
  Gut Microbiome composition and diversity will be assessed using 16 rRNA sequencing and Shotgun metagenomics in fecal samples collected in Shield Fecal Tubes, after 4 weeks of diet intervention

SECONDARY OUTCOMES:
Serum C-terminal telopeptide (CTX) | 4 weeks
  Serum Bone Turnover Marker C-terminal telopeptide (CTX) (ng/ml), will be assessed in fasting serum samples collected after 4 weeks of diet intervention
Proinflammatory Cytokines | 4 weeks
  Serum levels of Proinflammatory Cytokines: tumor necrosis factor α (TNFα), transforming growth factor beta (TGF beta) and interleukin-17 (IL-17) will be assessed in fasting serum samples collected after 4 weeks of diet intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ornit Cohen, Study Director — Wolfson Medical Center. Head of the Authority for Research and Innovation.; Rachel C Rosenblum, MD, Principal Investigator — Wolfson Medical Center. Endocrinology and Diabetes Unit; Orit Twito, MD, Study Chair — Wolfson Medical Center. Head of Endocrinology and Diabetes Unit